CLINICAL TRIAL: NCT03415477
Title: Denosumab: A Potential Treatment Option for Aneurysmal Bone Cysts
Acronym: Deno-ABC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Director, Head of Muscoloskeletal Tumor Center, Principal Investigator, Clinical Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Denosumab-ABC
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Bone Cyst Aneurysmal; Pathological Fracture; Recurrent Disease; Refractory Tumor
Keywords: aneurysmal bone cyst, denosumab, surgical treatment, complication
MeSH Terms: conditions — Bone Cysts, Aneurysmal; Fractures, Spontaneous; Recurrence; Neoplasms | interventions — Denosumab; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients with recurrent and/or refractory aneurysmal bone cysts treated with denosumab perioperatively.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- denosumab (Xgeva) treatment (Experimental): Patients with aneurismal bone cysts received perioperative denosumab(Xgeva).
  Interventions: Drug: Denosumab (Xgeva)

INTERVENTIONS:
Drug: Denosumab (Xgeva) — Denosumab (Xgeva) 120 mg was given subcutaneously (abdomen wall or upper arms) every 4 weeks (Q4W), with a loading dose on both Day 8 and Day15 of the first cycle， perioperatively.
  Other Names: surgical treatment

SUMMARY:
The efficacy of traditional therapeutic approaches for aneurysmal bone cysts (ABC), such as surgery, embolization, sclerotherapy and radiotherapy, are often compromised for lesions in axial skeletons and adolescents complicated with pathological fracture. Therefore, denosumab, a new drug that has been successfully used in giant cell tumor of bone but has seldom used in ABC, was used to treat ABC in this trial.

DETAILED DESCRIPTION:
Patients with primary ABC treated with perioperative denosumab in the Musculoskeletal Tumor Center of Peking University People's Hospital between January 2014 and December 2016 will be reported in this trial.Approved by the Ethics Committee of Peking University People's Hospital and with the full informed consent from the patients or their families, all patients received surgery and treatment with denosumab perioperatively. Denosumab 120 mg was given subcutaneously (abdomen wall or upper arms) every 4 weeks (Q4W), with a loading dose on both Day 8 and Day 15 of the first cycle. Meanwhile, all patients were suggested to take 800mg oral calcium supplement every day and avoid any dental or oral surgery (tooth extraction, tooth filling, etc.). Patients were followed once a month since the date of surgery. On follow-up visits, patient-reported adverse reactions, X-ray image of jawbone, serum calcium, alkaline phosphatase, renal and hepatic function, hemoglobin, white blood cell, and platelet count were collected, and histological examinations, radiological examinations (such as X-ray, computed tomography (CT), magnetic resonance image (MRI) and positron emission tomography-computed tomography (PET-CT) and postoperative functional status evaluations by MSTS（Musculoskeletal tumor society） score were conducted.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed with primary aneurysmal bone cyst
2. lesions in axial skeletons (i.e. spine, pelvis) which are difficult to reach a satisfactory surgical margin, and surgery can lead to very high incidence of complications.
3. pathological fracture
4. recurrence cases

Exclusion Criteria:

1. metastases or multi-focal lesions
2. malignancy

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | at least 1-year
  the number of participats (complete response+ partial response according to RECIST 1.1)/ total participants number.
local control rate | at least 1-year
  CT or MR proof that the tumor relapse in the primary site by at least two radiologist.

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory values and/or adverse events that are related to the use of Denosumab（Xgeva） | at least 1-year
  include patient-reported adverse reactions, X-ray image of jawbone, serum calcium, alkaline phosphatase, renal and hepatic function, hemoglobin, white blood cell, and platelet count were collected in follow-up every 3-month.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghermandi R, Terzi S, Gasbarrini A, Boriani S. Denosumab: non-surgical treatment option for selective arterial embolization resistant aneurysmal bone cyst of the spine and sacrum. Case report. Eur Rev Med Pharmacol Sci. 2016 Sep;20(17):3692-5. PMID 27649673
- [Background] Dubory A, Missenard G, Domont J, Court C. Interest of Denosumab for the Treatment of Giant-cells Tumors and Aneurysmal Bone Cysts of the Spine. About Nine Cases. Spine (Phila Pa 1976). 2016 Jun;41(11):E654-E660. doi: 10.1097/BRS.0000000000001350. PMID 27244112
- [Background] Skubitz KM, Peltola JC, Santos ER, Cheng EY. Response of Aneurysmal Bone Cyst to Denosumab. Spine (Phila Pa 1976). 2015 Nov;40(22):E1201-4. doi: 10.1097/BRS.0000000000001027. PMID 26730528
- [Background] Pauli C, Fuchs B, Pfirrmann C, Bridge JA, Hofer S, Bode B. Response of an aggressive periosteal aneurysmal bone cyst (ABC) of the radius to denosumab therapy. World J Surg Oncol. 2014 Jan 20;12:17. doi: 10.1186/1477-7819-12-17. PMID 24438319